CLINICAL TRIAL: NCT07390058
Title: ESTIMATION OF INCREASED SURGICAL DRAINAGE OUTPUT FOLLOWING THORACOLUMBAR SURGERY: DRAINAGE VOLUME PREDICTION SCORE
Brief Title: ESTIMATION OF INCREASED SURGICAL DRAINAGE OUTPUT FOLLOWING THORACOLUMBAR SURGERY
Status: Not yet recruiting | Type: Observational
Sponsor: AKİF BULUT (Other)
Responsible Party: Sponsor-Investigator, AKİF BULUT, Assistant Investigator, Uludag University
Organization: Uludag University (Other)
Other Study IDs: 2025-24/04
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Drainage; Spinal (Fusion) Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Increased total drainage: In the study, increased total drainage is defined as a total drainage amount of 317 ml or more at the end of the drainage termination day.
- Decreased total drainage: Decreased total drainage is defined as a total drainage amount of less than 317 ml at the end of the drainage termination day.

SUMMARY:
In a study involving neurosurgeons worldwide, it was reported that most surgeons preferred the use of drains (186, 80.5%) and subfascial drains (169, 73.2%), with 52.87% of surgeons discontinuing drains based on time and 27.7% based on drainage volume (Cabrera et al. 2025). While the Enhanced Recovery After Surgery (ERAS) protocol does not recommend routine wound drainage for short-segment lumbar fusion surgery (Evidence Level Moderate, Recommendation Strength), the timing of drainage termination is based on drainage output (if drainage is below 50 ml) or based on postoperative days (day 2) (Han et al., 2024; Smith et al., 2019). We believe that further studies are needed to determine which patient groups require drains preoperatively and how long drains should remain in place postoperatively. This study, which aims to predict the amount of drainage during the perioperative period, will attempt to predict both the selective use of drains and how long to wait before discontinuing drainage in patients with drains. Lumbar subcutaneous fat thickness, previously used as a predictor of surgical site infections, will be tested for the first time in our study to determine whether it is a predictor of drainage output.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 participated in the study.
* Patients who have undergone long segment spinal surgery (2 or more segments).

Exclusion Criteria:

* Patients with developing dural rupture,
* Patients under 18 or over 80 years of age,
* Patients undergoing revision surgery,
* Patients undergoing short segment spinal fusion,
* Patients using drains other than standard-volume closed suction drainage,
* Patients with missing data,
* Patients experiencing mechanical problems with the drain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study by Li et al. (2025) titled "Risk factors leading to increased postoperative drainage in patients undergoing spinal fusion surgery" (group with excessive drainage output 60%, group with low drainage output 40%) was referenced in calculating the sample size. Using the G-power 3.1.9.7 program, a Z test (Logistic regression) was performed. Assuming a 5% type I error (α), a 95% confidence level (1-α), and 0.95 power (1-β), the total sample size for high drainage output was 325 (Odds ratio (OR): 2.25). To ensure an equal number of patients in each group, 326 patients will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Total drainage volume | 10 days
  Total drainage volume until the drain is removed in patients with a thoracolumbar drain following surgery.

IPD SHARING:
Plan to Share IPD: Undecided